CLINICAL TRIAL: NCT00521638
Title: A Phase 1/2 Dose Escalation Study of TRU-015 in Subjects With Relapsed or Refractory B Cell Non-Hodgkin's Lymphoma
Brief Title: Study Evaluating TRU-015 in B-Cell Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Collaborators: Emergent Product Development Seattle LLC (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3206K2-104
Record Dates: First submitted 2007-08-24; First posted 2007-08-28 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Lymphoma, B-Cell
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — TRU-015 protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: TRU-015

INTERVENTIONS:
Biological: TRU-015 — Intravenous administration; 400 mg, 700 mg, or 1000 mg; 1x/week dosing for 4 weeks

SUMMARY:
This is a study to evaluate the safety and efficacy of TRU-015 in treatment of B-cell Non-Hodgkin's Lymphoma (NHL).

TRU-015 is also currently being evaluated in multiple clinical studies for the treatment of autoimmune disorders. Over 300 patients have received TRU-015 in these studies, and the data observed to date support its safety in patients with autoimmune disorders.

Safety of an escalating dose of 4 weekly infusions of TRU-015 will be evaluated in subjects with relapsed NHL (see inclusion criteria for subtypes).

Once a maximum tolerated dose (MTD) is confirmed or maximum dose to be studied is determined to be safe and well tolerated, an expanded cohort of subjects with relapsed follicular NHL will be evaluated for efficacy.

ELIGIBILITY:
Main Inclusion Criteria:

* Subjects with CD20-positive, B cell NHL who, after at least 2 prior therapies of probable clinical benefit, have relapsed or refractory disease. The following histologies may be included*: lymphoplasmacytic lymphoma (formerly known as lymphoplasmacytoid lymphoma), splenic marginal zone B cell lymphoma, extranodal marginal zone B cell lymphoma of mucosa-associated lymphoid tissue, nodal marginal zone B cell lymphoma, follicular lymphoma, mantle cell lymphoma, diffuse large-cell B cell lymphoma, and mediastinal large B cell lymphoma. Small lymphocytic lymphoma will be included if it is a primary diagnosis and if the lymphoma cells are < 5.0 x 109/L (5000/mm3) in the peripheral blood. *Subjects enrolled in the preliminary efficacy cohorts must have relapsed, refractory, or persistent follicular lymphoma (persistent disease defined as computed tomography (CT) positive for 3 months after last treatment), and must not have received anti-CD20 targeted therapy within 3 months of receiving the first dose of test article. Subjects may be considered eligible after a single therapy of probable clinical benefit, if no further standard effective treatment is available in the opinion of the investigator. Prior CD20 immunophenotyping of tumors to document B cell NHL is acceptable. If such prior documentation is not available, then the immunophenotype of the current disease must be documented by fine-needle aspirate or biopsy, or by circulating CD20-positive NHL cells from peripheral blood before administration of test article.
* At least 1 measurable lesion that is 1.5 cm in at least 1 dimension by CT or magnetic resonance imaging (MRI), in an area of no prior radiation therapy, or documented progression in an area that was previously irradiated.
* Recovery to baseline or grade 1 [according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 3.0] from all acute adverse effects of prior therapies (excluding alopecia).

Main Exclusion Criteria:

* Candidate for potentially curative therapy that is available to the subject, in the clinical opinion of the investigator.
* Diagnosis of chronic lymphocytic leukemia, Burkitt's lymphoma, primary effusion lymphoma, and/or precursor B cell lymphoblastic lymphoma.
* Prior treatments: radioimmunotherapy; allogeneic hematopoietic stem cell transplant (within 6 months of first dose of study drug); chemotherapy, cancer immunosuppressive therapy, growth factors (except erythropoietin), or investigational agents (within 4 weeks of first dose of study drug); major surgery not related to debulking surgical procedures (within 3 weeks of first dose of study drug).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Safety: physical examinations, laboratory tests, adverse events. Maximum Tolerated Dose: dose-limiting toxicities. Efficacy: disease response and progression status per International Response Criteria for NHL. | 9 months

SECONDARY OUTCOMES:
Objective response rate in subjects with relapsed follicular NHL. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (7):
- United States (7):
  - Duarte, California
  - San Diego, California
  - Chicago, Illinois
  - Boston, Massachusetts
  - St Louis, Missouri
  - Buffalo, New York
  - Cleveland, Ohio